CLINICAL TRIAL: NCT00303277
Title: Do HMG CoA Reductase Inhibitors Affect Abeta Levels?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Responsible Party: Elaine R. Peskind, MD, Professor, Director of Clinical Research, Mental Health Service, VA Puget Sound Health Care System/University of Washington School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 21974
Record Dates: First submitted 2006-03-14; First posted 2006-03-16 (Estimated); Last update posted 2010-04-13 (Estimated); Status verified 2010-04

CONDITIONS: Alzheimer's Disease; Aging
Keywords: Alzheimer's disease; beta-amyloid; statins
MeSH Terms: conditions — Alzheimer Disease; Plaque, Amyloid | interventions — Simvastatin; Pravastatin; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): simvastatin
  Interventions: Drug: simvastatin
- 2 (Active Comparator): pravastatin
  Interventions: Drug: pravastatin

INTERVENTIONS:
Drug: simvastatin — simvastatin 40 mg tablets once per day for 12 weeks
  Other Names: Zocor
  Arms: 1
Drug: pravastatin — pravastatin 80 mg tablets once per day for 12 weeks
  Other Names: Lipitor
  Arms: 2

SUMMARY:
Recent evidence suggests that there is a significant overlap between AD and cerebrovascular disease. In fact, AD and cerebrovascular disease may share some of the same risk factors, including hypercholesterolemia. In addition, studies have suggested that the HMG Co-A reductase inhibitor lipid-lowering agents, known as "statins," decrease the risk of AD by up to 70%; however, effects differed by specific statin use. This study will compare two statins, simvastatin (which crosses the blood brain barrier) and pravastatin (which does not), with respect to their ability to alter blood and cerebrospinal fluid (CSF) levels of AD and inflammatory markers. The primary aim of the proposed study is to determine whether there is a reduction in Abeta with statins and whether the ability of the statin to cross the blood-brain barrier will affect its ability to decrease Abeta. If it can be demonstrated that statins alter AD-associated biomarkers, this would have broad implications for the treatment and prevention of AD.

DETAILED DESCRIPTION:
Recent evidence suggests that there is a significant overlap between AD and cerebrovascular disease. In fact, AD and cerebrovascular disease may share some of the same risk factors, including hypercholesterolemia. In addition, studies have suggested that the HMG Co-A reductase inhibitor lipid-lowering agents, known as "statins," decrease the risk of AD by up to 70%; however, effects differed by specific statin use. This study will compare two statins, simvastatin (which crosses the blood brain barrier) and pravastatin (which does not), with respect to their ability to alter blood and cerebrospinal fluid (CSF) levels of AD and inflammatory markers. The primary aim of the proposed study is to determine whether there is a reduction in Abeta with statins and whether the lipophilicity of the statin will affect its ability to decrease Abeta. In addition, the proposal will determine statin effects on both peripheral and central inflammation and whether the lipophilicity of the statin will affect its ability to decrease inflammation. If it can be demonstrated that statins alter AD-associated biomarkers, this would have broad implications for the treatment and prevention of AD.

This study will be performed in 60 cognitively normal middle-aged and older persons with hypercholesterolemia (total cholesterol >200 and/or LDL>130), presumably persons that have a lipid-related increased risk of AD and in whom alterations of CSF Abeta can be interpreted.The differential effects of the two statins will be evaluated in a 12-week randomized treatment trial with 30 subjects in each group.

Prior to randomization and following 12 weeks of treatment with simvastatin or pravastatin, subjects will undergo CSF and blood collection. In the CSF, concentrations of Abeta 1-40, Abeta 1-42, soluble APP, tau, 24S-hydroxycholesterol, apoE, total cholesterol, F2-isoprostanes, glucose, protein, and cell count will be measured. In the blood, concentrations of total cholesterol, HDL, LDL, triglyceride, phospholipids, fatty acids, 24S-hydroxycholesterol, apoE, apoB, apoA1, Abeta 1-40, Abeta 1-42, F2-isoprostanes, C-reactive protein, fibrinogen, iron, homocysteine, and albumin will be measured. Plasma simvastatin and pravastatin concentrations will be measured at study completion. APOE genotyping will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Total cholesterol > 200, and/or LDL > 130
* No cognitive impairment
* Statin-naive for at least one year
* Women must not be pregnant, nursing, or planning to become pregnant

Exclusion Criteria:

* Back ailments which would hinder LP procedure
* Neurological disease, including stroke, Parkinson's disease, Multiple Sclerosis, uncontrolled epilepsy, history of severe head trauma
* Hepatic disease
* Renal insufficiency
* Unstable medical disease
* Severe pulmonary disease
* Severe cardiac disease
* Uncontrolled hypertension (greater than 160/90)
* Uncontrolled hyper/hypothyroidism
* History of blood clotting abnormalities or platelet abnormalities
* History of chronic major psychiatric disorders or presence of current major depressive disorder (by DSM-IV criteria)
* History of substance abuse within the past year
* Taking exclusionary medications

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2002-08; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
CSF abeta levels | baseline and 12 weeks

SECONDARY OUTCOMES:
CSF biomarkers | baseline and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elaine R Peskind, MD, Principal Investigator — University of Washington
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States

REFERENCES:
- [Background] Li G, Larson EB, Sonnen JA, Shofer JB, Petrie EC, Schantz A, Peskind ER, Raskind MA, Breitner JC, Montine TJ. Statin therapy is associated with reduced neuropathologic changes of Alzheimer disease. Neurology. 2007 Aug 28;69(9):878-85. doi: 10.1212/01.wnl.0000277657.95487.1c. PMID 17724290
- [Background] Li G, Higdon R, Kukull WA, Peskind E, Van Valen Moore K, Tsuang D, van Belle G, McCormick W, Bowen JD, Teri L, Schellenberg GD, Larson EB. Statin therapy and risk of dementia in the elderly: a community-based prospective cohort study. Neurology. 2004 Nov 9;63(9):1624-8. doi: 10.1212/01.wnl.0000142963.90204.58. PMID 15534246
- [Result] Riekse RG, Li G, Petrie EC, Leverenz JB, Vavrek D, Vuletic S, Albers JJ, Montine TJ, Lee VM, Lee M, Seubert P, Galasko D, Schellenberg GD, Hazzard WR, Peskind ER. Effect of statins on Alzheimer's disease biomarkers in cerebrospinal fluid. J Alzheimers Dis. 2006 Dec;10(4):399-406. doi: 10.3233/jad-2006-10408. PMID 17183151